CLINICAL TRIAL: NCT02341235
Title: Self-monitoring Activity: a Randomized Trial of Game-oriented Applications (SMARTGOAL)
Brief Title: Self-monitoring Activity: a Randomized Trial of Game-oriented Applications
Acronym: SMARTGOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-0376
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Obesity
Keywords: video game; narrative; story; survivorship; cancer survivor; mhealth; physical activity; women; women's health
MeSH Terms: conditions — Breast Neoplasms; Obesity; Narration; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Game intervention (Experimental): Participants will receive narrative-based games on a mobile device and telephone counseling (weekly for the first 12 weeks, then once per month until 6 months)
  Interventions: Behavioral: Game intervention
- Standard intervention (Active Comparator): Participants will receive an electronic activity monitor with a mobile device and telephone counseling (weekly for the first 12 weeks, then once per month until 6 months)
  Interventions: Behavioral: Standard intervention

INTERVENTIONS:
Behavioral: Game intervention — The game will target motivation via narrative and game mechanics. It will also encourage self-regulation by providing monitoring and feedback of activity. Counseling will be adapted to specifically reference concepts related to narrative and games.
  Arms: Game intervention
Behavioral: Standard intervention — The electronic activity monitor will monitor steps, and the mobile device will provide basic feedback on progress toward goals. Counseling will be standard and concentrate on self-regulatory skill-building.
  Arms: Standard intervention

SUMMARY:
The purpose of this study is to compare an enhanced intervention that includes narrative and game components to a standard intervention that only targets self-monitoring. These approaches will be tested among postmenopausal breast cancer survivors who are sedentary and overweight.

DETAILED DESCRIPTION:
Habitual physical activity decreases risk of multiple negative health outcomes, including breast cancer recurrence and mortality. It is also associated with better quality of life and reducing negative effects of cancer and cancer treatment. However, most breast cancer survivors do not engage in sufficient physical activity. Behavior change interventions produce short-term increases in activity but have difficulty motivating sustained active lifestyles over longer periods and are not equally effective in women of different races/ethnicities. The purpose of this study is to test a novel intervention that uses video games and storytelling to increase motivation. Video game mechanics increase enjoyment and feelings of autonomy (control), competence, and relatedness to others. All of these feelings are associated with motivation for activity and, in turn, sustained activity over time. Additionally, narrative storytelling is an effective method of persuading individuals to change their behavior. We propose that play of active video games that include compelling storylines will increase physical activity among a diverse sample of postmenopausal breast cancer survivors.

To test this hypothesis, we will conduct a clinical trial that compares the enhanced intervention (story-based video games) to a standard intervention in 90 sedentary, overweight postmenopausal breast cancer survivors. Participants in the enhanced group will receive a mobile device and accessories with two story-based video game applications installed. The games incorporate behavior change strategies such as self-monitoring and feedback while also using game mechanics and a lengthy storyline to motivate physical activity. Participants in the standard group will receive the same mobile device with an electronic activity monitor and its companion feedback application. Both groups will receive brief weekly telephone counseling. By comparing two groups that both receive typical behavior change intervention components (counseling) and a novel electronic intervention, we will be able to investigate the specific effects of game mechanics and storytelling on motivation and physical activity. We will measure changes in physical activity, fitness, function, and quality of life from the beginning of the study to 6 months. We will also investigate further changes during an additional 6 month follow-up period in which participants keep their intervention tools but do not receive any counseling, to measure maintenance of activity. This project will develop and test a promising, innovative intervention that has the potential to be used on a widespread basis in clinical and community settings.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 45 and 75 years old
2. Report a breast cancer diagnosis no more than 10 years prior to enrollment
3. Cessation of menses for 12 months or more
4. Able to read and understand English
5. Able to read words in standard applications on a mobile device 3-4" large
6. Able to walk for exercise
7. Able to find transportation to the study location
8. Willing to use a mobile device provided by the study to participate (or to use one of their own)
9. Willing to be randomized to either group

Exclusion Criteria:

1. Currently pregnant or nursing
2. Surgery in the past six months
3. Chemotherapy or radiation treatment in the past six months
4. Evidence of disease recurrence
5. Participant is active (90 minutes of moderate-vigorous intensity activity per week or more)
6. BMI is under 25 kg/m2 or over 35 kg/m2
7. Report a heart condition, chest pain during periods of activity or rest, loss of consciousness, etc. on the Physical Activity Readiness Questionnaire (PAR-Q), unless cleared by their physician
8. Participant reports hospitalization within the past year due to psychiatric problem(s)
9. Report current symptoms of alcohol or substance dependence
10. Plans to move away from the Galveston-Houston area or to be out of town for more than 1 week during the study period
11. Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
12. Report a history of severe orthopedic complications that would prevent optimal participation in the physical activities prescribed (e.g., severe arthritis, leg amputations, etc.)
13. Clinical judgment concerning safety
14. Lost more than 5% body weight in the previous 6 months
15. Currently participating in a physical activity or weight loss program
16. Current smoker
17. Participant already uses an electronic activity monitor (we will ask them to stop)
18. Another member of the household is a participant or staff member on this trial

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Lyons EJ, Baranowski T, Basen-Engquist KM, Lewis ZH, Swartz MC, Jennings K, Volpi E. Testing the effects of narrative and play on physical activity among breast cancer survivors using mobile apps: study protocol for a randomized controlled trial. BMC Cancer. 2016 Mar 9;16:202. doi: 10.1186/s12885-016-2244-y. PMID 26960972

RESULTS

PARTICIPANT FLOW:
Period: Baseline to 6 Months
Arm/Group | Game Intervention | Standard Intervention
Started | 45 | 45
Completed | 28 | 31
Not Completed | 17 | 14
Period: 6 Months to 12 Months
Arm/Group | Game Intervention | Standard Intervention
Started | 28 | 31
Completed | 22 | 21
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Game Intervention | Standard Intervention | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.48 (6.78) | 59.92 (7.68) | 61.22 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 39 | 40 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 37 | 33 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Time since diagnosis [Mean (Standard Deviation); unit: years] | 5.55 (6.43) | 6.84 (5.29) | 6.19 (5.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in Minutes Per Day of Physical Activity
Description: Minutes of moderate-vigorous physical activity per day (averaged over a 7 day period) at baseline and 6 months.
Time Frame: baseline and 6 months
Measure: Mean (Standard Error); unit: minutes per day
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
minutes per day | 20.87 (3.29) | 15.82 (3.54)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .35, ANCOVA

2. Secondary Outcome: Change in Physical Fitness From Baseline to 6 Months, as Measured by 6 Minute Walk Test
Description: We will use a 6 minute walk test to measure fitness, measured in feet walked in six minutes on a pre-marked indoor course
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: feet
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
feet | -44.35 (106.92) | 71.74 (88.64)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = 0.22, ANCOVA

3. Secondary Outcome: Change in Physical Function From Baseline to 6 Months as Measured by the Senior Fitness Test's Chair Stand Measure
Description: We will use the Senior Fitness Test to measure physical function, specifically in regards to the number of chair stands that can be completed within 30 seconds. A higher number indicates better function in this area.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: number of chair stands
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
number of chair stands | .33 (1.35) | .4 (1.02)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .97, ANCOVA

4. Secondary Outcome: Change in Weight From Baseline to 6 Months
Description: We will measure weight using a calibrated scale
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
pounds | -.14 (4.37) | -.04 (2.94)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .98, ANCOVA

5. Secondary Outcome: Change in Physical Quality of Life From Baseline to 6 Months as Measured by Functional Assessment of Cancer Therapy - Breast Measure
Description: We will use the Functional Assessment of Cancer Therapy - Breast measure's physical subscale. This scale has a range of 0-28 and 7 items measured on a 5 point scale (not at all to very much). A higher score indicates greater physical quality of life.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | -1.11 (.93) | -1.39 (.88)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .83, ANCOVA

6. Secondary Outcome: Change in Intrinsic Motivation From Baseline to 6 Months, Measured by Intrinsic Motivation Specific to Physical Activity
Description: The Behavioral Regulation in Exercise Questionnaire-2 intrinsic regulation subscale will be used. This subscale includes 4 items measured using a 5 point scale (not true for me to very true for me), with a range of scores from 0-12. A higher number indicates higher intrinsic motivation.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | .11 (.23) | .62 (.22)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .055, ANCOVA

7. Secondary Outcome: Change in Social/Family Quality of Life From Baseline to 6 Months as Measured by Functional Assessment of Cancer Therapy - Breast Measure's Social/Family Well-Being Subscale
Description: We will use the Functional Assessment of Cancer Therapy - Breast measure's social/family subscale. This scale has a range of 0-28 and 7 items measured on a 5-point scale (not at all to very much). A higher score indicates greater social/family quality of life.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | -.74 (1.27) | -1.53 (1.11)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .71, ANCOVA

8. Secondary Outcome: Change in Emotional Quality of Life From Baseline to 6 Months as Measured by Functional Assessment of Cancer Therapy - Breast Measure's Emotional Well-Being Subscale
Description: We will use the Functional Assessment of Cancer Therapy - Breast measure's emotional subscale. This scale has a range of 0-24 and 6 items measured on a 5-point scale (not at all to very much). A higher score indicates greater emotional quality of life
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | -1.76 (1.16) | -.27 (.95)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .33, ANCOVA

9. Secondary Outcome: Change in Functional Quality of Life From Baseline to 6 Months as Measured by Functional Assessment of Cancer Therapy - Breast Measure's Functional Well-Being Subscale
Description: We will use the Functional Assessment of Cancer Therapy - Breast measure's functional subscale. This scale has a range of 0-28 and 7 items measured on a 5-point scale (not at all to very much). A higher score indicates greater functional quality of life
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | .72 (1.14) | .6 (.87)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .94, ANCOVA

10. Secondary Outcome: Change in Breast Cancer-Specific Quality of Life From Baseline to 6 Months as Measured by Functional Assessment of Cancer Therapy - Breast Measure's Breast Cancer Subscale
Description: We will use the Functional Assessment of Cancer Therapy - Breast measure's breast cancer subscale. This scale has a range of 0-40 and 10 items measured on a 5-point scale (not at all to very much). A higher score indicates greater breast cancer-related quality of life
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | -0.03 (1.16) | -.96 (1.34)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .57, ANCOVA

11. Secondary Outcome: Change in Identified Regulation From Baseline to 6 Months, Measured by Identified Regulation Specific to Physical Activity
Description: The Behavioral Regulation in Exercise Questionnaire-2 identified regulation subscale will be used. This subscale includes 4 items measured using a 5 point scale (not true for me to very true for me), with a range of scores from 0-12. A higher number indicates a greater amount of identified regulation.
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | .01 (.19) | .30 (.21)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .30, ANCOVA

12. Secondary Outcome: Change in Integrated Regulation From Baseline to 6 Months, Measured by Integrated Regulation Specific to Physical Activity
Description: We will use items from P.M. Wilson and colleague's expansion of the Behavioral Regulation in Exercise Questionnaire-2 to include integrated regulation. This subscale includes 4 items measured using a 5 point scale (not true for me to very true for me), with a range of scores from 0-12. A higher number indicates a greater amount of identified regulation.
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
units on a scale | .32 (.27) | .53 (.18)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .44, ANCOVA

13. Secondary Outcome: Change in Physical Function From Baseline to 6 Months as Measured by the Senior Fitness Test's Arm Curl Measure
Description: We will use the Senior Fitness Test to measure physical function, specifically in regards to the number of arm curls that can be completed within 30 seconds. A higher number indicates better function in this area.
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: number of arm curls
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
number of arm curls | .39 (1.34) | 1.04 (.83)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .62, ANCOVA

14. Secondary Outcome: Change in Physical Function From Baseline to 6 Months as Measured by the Senior Fitness Test's Sit and Reach Measure
Description: We will use the Senior Fitness Test to measure physical function, specifically in regards to the distance an individual can reach from their toes when bending forward. A higher number indicates better function in this area.
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: inches
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
inches | -.05 (.73) | .29 (.63)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .70, ANCOVA

15. Secondary Outcome: Change in Physical Function From Baseline to 6 Months as Measured by the Senior Fitness Test's Back Scratch Measure
Description: We will use the Senior Fitness Test to measure physical function, specifically in regards to the distance between an individual's arms when they reach them behind their back (one higher above the shoulder and one lower). A higher number indicates better function in this area.
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: inches
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
inches | 1.32 (1.98) | -.57 (.91)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .41, ANCOVA

16. Secondary Outcome: Change in Physical Function From Baseline to 6 Months as Measured by the Senior Fitness Test's 8 Foot Up and Go Test
Description: We will use the Senior Fitness Test to measure physical function, specifically in regards to the time in which an individual can sit up, walk 8 feet around a cone, and sit back down. A lower number indicates better function in this area.
Time Frame: baseline to 6 Months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
seconds | .68 (.85) | .26 (.85)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; All analyses were adjusted for baseline values, age, race, ethnicity, and time since diagnosis; Test type: Superiority; p = .72, ANCOVA

17. Other Pre Specified Outcome: Maintenance of Physical Fitness From 6 Months to 1 Year, Measured by a 6 Minute Walk Test
Description: as for outcome 2
Time Frame: baseline to 6 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Maintenance of Physical Function From 6 Months to 1 Year, Measured by the Senior Fitness Test
Description: We will use the Senior Fitness Test to measure physical function, with a higher number indicating greater function
Time Frame: baseline to 6 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Sleep From 6 Months to 1 Year
Description: We will use a computerized PROMIS measure specific to cancer survivors
Time Frame: baseline to 6 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Weight From 6 Months to 1 Year
Description: Weight will be measured using a calibrated scale
Time Frame: baseline to 6 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Adherence, Measured by Objective Measures to Investigate Adherence to Study Protocols
Description: We will use objective measures to investigate adherence to study protocols (game usage, monitor usage, phone calls completed, assessments attended, etc.)
Time Frame: 1 year
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Number of Participants Who Report Adverse Events
Description: We will inquire about potential adverse events during counseling calls and assessment visits. Discrete events will be summed, and the number of participants with events will be summed.
Time Frame: 1 year
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Change in Anxiety From Baseline to 6 Months
Description: We will use a computerized PROMIS measure to investigate anxiety (Patient Reported Outcomes Measurement Information System PROMIS-Ca Bank 1.0 - Anxiety). The result shown is a t-score, where a score of 50 would be equivalent to the mean in the population of cancer survivors. Because the standard deviation is 10, a score of 10 higher or lower would indicate that the score is 1 standard deviation higher or lower (more/less anxiety) than the population.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
t-score | 51.34 (0.90) | 49.09 (0.90)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; Test type: Superiority; p = 0.084, ANCOVA

24. Other Pre Specified Outcome: Change in Depression From 6 Months to 1 Year
Description: We will use a computerized PROMIS measure specific to cancer patients/survivors (Patient Reported Outcomes Measurement Information System PROMIS-Ca Bank 1.0 - Depression)
Time Frame: baseline to 6 months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in Fatigue From Baseline to 6 Months
Description: We will use a computerized PROMIS measure specific to cancer patients/survivors (Patient Reported Outcomes Measurement Information System PROMIS-Ca Bank 1.0 Fatigue). The result shown is a t-score, where a score of 50 would be equivalent to the mean in the population of cancer survivors. Because the standard deviation is 10, a score of 10 higher or lower would indicate that the score is 1 standard deviation higher or lower (more/less fatigued) than the population.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
t-score | 50.96 (0.75) | 50.37 (0.75)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; Test type: Superiority; p = 0.580, ANCOVA

26. Other Pre Specified Outcome: Change in Quality of Life From 6 Months to 1 Year
Description: We will use the Functional Assessment of Cancer Therapy - Breast measure
Time Frame: baseline to 6 months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Change in Motivation From 6 Months to 1 Year, Measured by Autonomous Motivation Specific to Physical Activity
Description: Behavioral Regulation in Exercise Questionnaire-2 will be used, specifically subscales for autonomous motivation (intrinsic, integrated, identified regulation). We will use items from P.M. Wilson and colleague's expansion of the Behavioral Regulation in Exercise Questionnaire-2 to include integrated regulation.
Time Frame: baseline to 6 months
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Acceptability, Measured Using Self-report Measures of Usability and Liking of the Apps
Description: Participants will report their perceptions of app usability and acceptability in the 6 month questionnaire
Time Frame: baseline to 6 months
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Play Experience, Measured Using the Play Experience Questionnaire
Description: Participants will self-report their perceptions of the playfulness of the intervention apps
Time Frame: Measured at 3 months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Change in Exercise Identity From Baseline to 6 Months
Description: We will use the Exercise Identity Scale to investigate exercise beliefs and exercise role identity
Time Frame: baseline to 6 months
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Narrative Engagement (Measured in Narrative Group Only), Measured Using the Narrative Engagement Scale
Description: We will measure the extent to which participants in the narrative group felt narratively engaged in the game's storyline
Time Frame: Measured at 3 months
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Character Identification (Measured in Narrative Group Only), Measured Using the Player Identification Scale
Description: We will measure the extent to which participants in the narrative group felt like they identified with their game character
Time Frame: Measured at 3 months
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Change in Depression From Baseline to 6 Months
Description: We will use a computerized PROMIS measure specific to cancer patients/survivors (Patient Reported Outcomes Measurement Information System PROMIS-Ca Bank 1.0 - Depression). The result shown is a t-score, where a score of 50 would be equivalent to the mean in the population of cancer survivors. Because the standard deviation is 10, a score of 10 higher or lower would indicate that the score is 1 standard deviation higher or lower (more/less depressed) than the population.
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
t-score | 49.32 (0.77) | 48.50 (0.77)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; Test type: Superiority; p = 0.461, ANCOVA

34. Other Pre Specified Outcome: Change in Fatigue From 6 Months to 1 Year
Description: We will use a computerized PROMIS measure specific to cancer patients/survivors
Time Frame: baseline to 6 months
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change in Sleep From Baseline to 6 Months
Description: We will use a computerized PROMIS measure (Patient Reported Outcomes Measurement Information System PROMIS Bank v1.0 - Sleep-Related Impairment). The result shown is a t-score, where a score of 50 would be equivalent to the mean in the population. Because the standard deviation is 10, a score of 10 higher or lower would indicate that the score is 1 standard deviation higher or lower than the population (more/less impairment).
Time Frame: baseline to 6 months
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Game Intervention | Standard Intervention
Number analyzed (Participants) | 45 | 45
t-score | 52.35 (0.48) | 52.30 (0.48)
Statistical Analysis 1: Comparison: Game Intervention vs Standard Intervention; Test type: Superiority; p = 0.934, ANCOVA

36. Other Pre Specified Outcome: Maintenance of Physical Activity From 6 Months to 1 Year
Description: Minutes of moderate-vigorous physical activity measured over a 7 day period
Time Frame: baseline to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Game Intervention | Standard Intervention
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/45 | 2/45
Other Adverse Events (participants affected / at risk) | 3/45 | 2/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Game Intervention (N=45) | Standard Intervention (N=45)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Gastroenteritis
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Breast reconstruction surgery
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) — Chest pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Game Intervention (N=45) | Standard Intervention (N=45)
Back pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Broken toe (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Achilles tendon tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Please interpret numerical outcomes with caution due to large amounts of drop out and low adherence in this pilot trial. All pre-specified PROMIS outcomes that were collected are provided, but note that these measures in particular faced a large amount of missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT02341235/Prot_SAP_000.pdf